CLINICAL TRIAL: NCT02931968
Title: A Retrospective Clinical Study Evaluating Full-Arch Monolithic Zirconia Implant Supported Fixed Dental Prosthesis
Brief Title: Full-arch Monolithic Zirconia ISFDP Follow up
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: 16-0550
Record Dates: First submitted 2016-10-11; First posted 2016-10-13 (Estimated); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Edentulous
Keywords: Monolithic Zirconia; Implant supported prosthesis; Fixed partial denture
MeSH Terms: conditions — Mouth, Edentulous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Monolithic zirconia prosthesis: Subjects previously treated with at least one arch (maxilla/mandible) of dental implants restored with a full-arch monolithic zirconia implant supported fixed dental prosthesis will be recalled for clinical and radiographic examination.
  Interventions: Device: Monolithic zirconia prosthesis

INTERVENTIONS:
Device: Monolithic zirconia prosthesis — Edentulous arch subjects treated with a monolithic zirconia implant supported fixed dental prosthesis.

SUMMARY:
This study is designed to recall all patients who have received a full-arch monolithic zirconia implant supported fixed dental prosthesis in the University of North Carolina (UNC) School of Dentistry Graduate Prosthodontic and/or Dental Faculty Practice clinics between January 1, 2008 to September 1, 2015. The main purpose is to evaluate the biological and technical complications associated with this form of prosthetic treatment. Additionally patient centered outcomes will be evaluated.

DETAILED DESCRIPTION:
Purpose: A retrospective single-center study to provide scientific data on the clinical performance of full-arch monolithic zirconia implant supported fixed dental prosthesis (MZISFDP).

Participants: Individuals with at least one edentulous dental arch (maxilla/mandible) who were treated in the UNC Graduate Prosthodontic clinic and Dental Faculty Practice between January 1, 2008 to September 1, 2015 with full-arch MZISFDP.

Procedures (methods): This study is designed as a retrospective descriptive study with a single prospective examination of a population of subjects previously restored with full-arch MZISFDPs. An estimated 60 participants will be enrolled in the study. The study includes retrospective data and radiograph collection from dental records as well as data collection from one prospective visit that includes clinical examination, a panoramic radiograph and 2 patient questionnaires.

ELIGIBILITY:
Inclusion Criteria

* 18 years and older
* Good physical health (American Society of Anesthesiologist classification I (ASA I) and II (ASA II) to undergo routine comprehensive recall examination

  1. ASA I - A normal healthy patient
  2. ASA II - A patient with mild systemic health.
* Able to give informed consent
* At least one edentulous arch (maxilla and/or mandible) that were treatment planned and restored with full arch MZISFDP by UNC Graduate Prosthodontic clinic and/or UNC Dental Faculty Practice between January 1, 2008- September 1, 2015
* Pregnancy status during the time of recall

  1. Women of non-childbearing potential - defined as those who have no uterus, ligation of the fallopian tubes, or permanent cessation of ovarian function due to ovarian failure or surgical removal of the ovaries (i.e. permanently sterilized, postmenopausal). Postmenopausal is defined as 12 months with no menses without an alternative medical cause "Non-childbearing potential" status will be determined with a questionnaire.
  2. Women of childbearing potential - Female patient who don't fulfill the "non-childbearing potential" status will be considered of childbearing potential. Status of pregnancy will be determined by administering urine pregnancy tests If a subject is found to be pregnant and they consent to remaining in the study then any data from the intraoral exam will be included and the subject will be excluded from the radiographic examination.

Exclusion Criteria

* History of radiotherapy in the head and neck region
* History of intravenous bisphosphonate therapy
* Medical conditions that contraindicate elective dental therapy and routine recall appointment
* American Society of Anesthesiologist Classification III (ASA III), IV (ASA IV), V (ASA V) and VI (ASA VI)

  1. ASA III - a patient with severe systemic disease
  2. ASA IV -a patient with severe systemic disease that is a constant threat to life.
  3. ASA V - a moribund patient who is not expected to survive without the operation.
  4. ASA VI - a declared brain-dead patient whose organs are being removed for donor purposes.
* Psychological and/or behavioral conditions that make routine recall appointments very difficult to impossible
* Known alcohol and/or drug abuse

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adult patients treated in the UNC School of Dentistry Graduate Prosthodontic and/or Dental Faculty Practice clinic(s) between January 1, 2008 to September 1, 2015 with at least one full-arch monolithic zirconia implant supported fixed dental prosthesis.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-11-05 (Actual); Study Completion 2018-11-05 (Actual)

PRIMARY OUTCOMES:
Percent Incidence of Prosthetic Complications | At time of study visit (anywhere from 1-8 years from prosthesis delivery)
  Implant and prosthetic survivals are going to be reported by number of occurrence and will be analyzed by using descriptive tabular methods; Prosthetic screw loosening (number of complications calculated by percent), Repair of prosthesis (zirconia fracture)

SECONDARY OUTCOMES:
Percent Incidence of Biological Complications | At time of study visit (anywhere from 1-8 years from prosthesis delivery)
  Biological complications are going to be reported by number of sites and mm around bone loss and will be analyzed by using descriptive tabular methods; Bleeding on probing, Bone loss around implant fixture
Quantitative measurement of bone level | At time of study visit (anywhere from 1-8 years from prosthesis delivery)
  A standard panoramic radiograph will be obtained to assess hard tissue status around each dental implant supporting the prosthesis, which will be measured by using a software program.
Patient self-reported OHIP-14 satisfaction scores | At time of study visit (anywhere from 1-8 years from prosthesis delivery)
  Oral Health Impact Profile 14 (OHIP-14) will be administered to evaluate patient centered outcomes with regards to prosthesis. Responses are organized into 5 subscales (not at all satisfied, not very satisfied, reasonably satisfied, very satisfied, totally satisfied) and are based on a Likert scale.
Patient self-reported QoLFAST-10 scores | At time of study visit (anywhere from 1-8 years from prosthesis delivery)
  Patient paper questionnaire; Quality of life related to function, aesthetics, socialization, and thoughts about health-behavioral habits (QoLFAST-10) will be administered to evaluate patient centered outcomes with regards to prosthesis. Responses are organized into 5 subscales (strongly disagree, disagree, indifferent, agree, strongly agree) and are based on a Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Ingeborg De Kok, DDS MS, Principal Investigator — UNC Associate Professor
Locations (1):
- Graduate Prosthodontic Clinic, Dept. of Prosthodontics, UNC School of Dentistry, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdulmajeed AA, Lim KG, Narhi TO, Cooper LF. Complete-arch implant-supported monolithic zirconia fixed dental prostheses: A systematic review. J Prosthet Dent. 2016 Jun;115(6):672-677.e1. doi: 10.1016/j.prosdent.2015.08.025. Epub 2016 Jan 23. PMID 26809220
- [Background] Al-Amleh B, Lyons K, Swain M. Clinical trials in zirconia: a systematic review. J Oral Rehabil. 2010 Aug;37(8):641-52. doi: 10.1111/j.1365-2842.2010.02094.x. Epub 2010 Apr 9. PMID 20406352
- [Background] Allen F, McMillan A. Food selection and perceptions of chewing ability following provision of implant and conventional prostheses in complete denture wearers. Clin Oral Implants Res. 2002 Jun;13(3):320-6. doi: 10.1034/j.1600-0501.2002.130313.x. PMID 12010164
- [Background] Attard NJ, Zarb GA. Long-term treatment outcomes in edentulous patients with implant-fixed prostheses: the Toronto study. Int J Prosthodont. 2004 Jul-Aug;17(4):417-24. PMID 15382777
- [Background] Balshi TJ, Wolfinger GJ, Slauch RW, Balshi SF. A retrospective analysis of 800 Branemark System implants following the All-on-Four protocol. J Prosthodont. 2014 Feb;23(2):83-8. doi: 10.1111/jopr.12089. Epub 2013 Jul 25. PMID 23890014
- [Background] Bozini T, Petridis H, Garefis K, Garefis P. A meta-analysis of prosthodontic complication rates of implant-supported fixed dental prostheses in edentulous patients after an observation period of at least 5 years. Int J Oral Maxillofac Implants. 2011 Mar-Apr;26(2):304-18. PMID 21483883
- [Background] Carames J, Tovar Suinaga L, Yu YC, Perez A, Kang M. Clinical Advantages and Limitations of Monolithic Zirconia Restorations Full Arch Implant Supported Reconstruction: Case Series. Int J Dent. 2015;2015:392496. doi: 10.1155/2015/392496. Epub 2015 Jun 1. PMID 26124835
- [Background] Cheng CW, Chien CH, Chen CJ, Papaspyridakos P. Complete-mouth implant rehabilitation with modified monolithic zirconia implant-supported fixed dental prostheses and an immediate-loading protocol: a clinical report. J Prosthet Dent. 2013 Jun;109(6):347-52. doi: 10.1016/S0022-3913(13)00109-1. No abstract available. PMID 23763777
- [Background] Cooper LF. The current and future treatment of edentulism. J Prosthodont. 2009 Feb;18(2):116-22. doi: 10.1111/j.1532-849X.2009.00441.x. PMID 19254301
- [Background] Davis DM, Packer ME, Watson RM. Maintenance requirements of implant-supported fixed prostheses opposed by implant-supported fixed prostheses, natural teeth, or complete dentures: a 5-year retrospective study. Int J Prosthodont. 2003 Sep-Oct;16(5):521-3. PMID 14651238
- [Background] de Avila ED, Avila-Campos MJ, Vergani CE, Spolidorio DM, Mollo Fde A Jr. Structural and quantitative analysis of a mature anaerobic biofilm on different implant abutment surfaces. J Prosthet Dent. 2016 Apr;115(4):428-36. doi: 10.1016/j.prosdent.2015.09.016. Epub 2015 Nov 17. PMID 26597465
- [Background] Douglass CW, Shih A, Ostry L. Will there be a need for complete dentures in the United States in 2020? J Prosthet Dent. 2002 Jan;87(1):5-8. doi: 10.1067/mpr.2002.121203. PMID 11807476
- [Background] Ekelund JA, Lindquist LW, Carlsson GE, Jemt T. Implant treatment in the edentulous mandible: a prospective study on Branemark system implants over more than 20 years. Int J Prosthodont. 2003 Nov-Dec;16(6):602-8. PMID 14714838
- [Background] Felton DA. Edentulism and comorbid factors. Tex Dent J. 2010 Apr;127(4):389-401. PMID 20446489
- [Background] Fueki K, Kimoto K, Ogawa T, Garrett NR. Effect of implant-supported or retained dentures on masticatory performance: a systematic review. J Prosthet Dent. 2007 Dec;98(6):470-7. doi: 10.1016/S0022-3913(07)60147-4. PMID 18061741
- [Background] Guess PC, Schultheis S, Bonfante EA, Coelho PG, Ferencz JL, Silva NR. All-ceramic systems: laboratory and clinical performance. Dent Clin North Am. 2011 Apr;55(2):333-52, ix. doi: 10.1016/j.cden.2011.01.005. Epub 2011 Mar 3. PMID 21473997
- [Background] Jemt T, Johansson J. Implant treatment in the edentulous maxillae: a 15-year follow-up study on 76 consecutive patients provided with fixed prostheses. Clin Implant Dent Relat Res. 2006;8(2):61-9. doi: 10.1111/j.1708-8208.2006.00003.x. PMID 16774591
- [Background] Kordatzis K, Wright PS, Meijer HJ. Posterior mandibular residual ridge resorption in patients with conventional dentures and implant overdentures. Int J Oral Maxillofac Implants. 2003 May-Jun;18(3):447-52. PMID 12814322
- [Background] Kwon T, Bain PA, Levin L. Systematic review of short- (5-10 years) and long-term (10 years or more) survival and success of full-arch fixed dental hybrid prostheses and supporting implants. J Dent. 2014 Oct;42(10):1228-41. doi: 10.1016/j.jdent.2014.05.016. Epub 2014 Jun 26. PMID 24975989
- [Background] Larsson C, Vult von Steyern P. Five-year follow-up of implant-supported Y-TZP and ZTA fixed dental prostheses. A randomized, prospective clinical trial comparing two different material systems. Int J Prosthodont. 2010 Nov-Dec;23(6):555-61. PMID 21209993
- [Background] Larsson C, Vult Von Steyern P. Implant-supported full-arch zirconia-based mandibular fixed dental prostheses. Eight-year results from a clinical pilot study. Acta Odontol Scand. 2013 Sep;71(5):1118-22. doi: 10.3109/00016357.2012.749518. Epub 2012 Dec 4. PMID 23210793
- [Background] Le M, Papia E, Larsson C. The clinical success of tooth- and implant-supported zirconia-based fixed dental prostheses. A systematic review. J Oral Rehabil. 2015 Jun;42(6):467-80. doi: 10.1111/joor.12272. Epub 2015 Jan 10. PMID 25580846
- [Background] Limmer B, Sanders AE, Reside G, Cooper LF. Complications and patient-centered outcomes with an implant-supported monolithic zirconia fixed dental prosthesis: 1 year results. J Prosthodont. 2014 Jun;23(4):267-75. doi: 10.1111/jopr.12110. Epub 2014 Jan 6. PMID 24393461
- [Background] Lund JP, Mojon P, Pho M, Feine JS. Alzheimer's disease and edentulism. Age Ageing. 2003 Mar;32(2):228-9. doi: 10.1093/ageing/32.2.228. No abstract available. PMID 12615571
- [Background] MacEntee MI, Nolan A, Thomason JM. Oral mucosal and osseous disorders in frail elders. Gerodontology. 2004 Jun;21(2):78-84. doi: 10.1111/j.1741-2358.2004.00008.x. PMID 15185987
- [Background] Mehra M, Vahidi F. Complete mouth implant rehabilitation with a zirconia ceramic system: a clinical report. J Prosthet Dent. 2014 Jul;112(1):1-4. doi: 10.1016/j.prosdent.2013.12.016. Epub 2014 Mar 24. PMID 24674807
- [Background] Mertens C, Steveling HG. Early and immediate loading of titanium implants with fluoride-modified surfaces: results of 5-year prospective study. Clin Oral Implants Res. 2011 Dec;22(12):1354-60. doi: 10.1111/j.1600-0501.2010.02123.x. Epub 2011 Mar 8. PMID 21382092
- [Background] Nascimento CD, Pita MS, Fernandes FHNC, Pedrazzi V, de Albuquerque Junior RF, Ribeiro RF. Bacterial adhesion on the titanium and zirconia abutment surfaces. Clin Oral Implants Res. 2014 Mar;25(3):337-343. doi: 10.1111/clr.12093. Epub 2013 Jan 14. PMID 23316996
- [Background] Oh SH, Kim Y, Park JY, Jung YJ, Kim SK, Park SY. Comparison of fixed implant-supported prostheses, removable implant-supported prostheses, and complete dentures: patient satisfaction and oral health-related quality of life. Clin Oral Implants Res. 2016 Feb;27(2):e31-7. doi: 10.1111/clr.12514. Epub 2014 Oct 24. PMID 25346286
- [Background] Papaspyridakos P, Chen CJ, Chuang SK, Weber HP, Gallucci GO. A systematic review of biologic and technical complications with fixed implant rehabilitations for edentulous patients. Int J Oral Maxillofac Implants. 2012 Jan-Feb;27(1):102-10. PMID 22299086
- [Background] Papaspyridakos P, Lal K. Complete arch implant rehabilitation using subtractive rapid prototyping and porcelain fused to zirconia prosthesis: a clinical report. J Prosthet Dent. 2008 Sep;100(3):165-72. doi: 10.1016/S0022-3913(08)00110-8. PMID 18762028
- [Background] Papaspyridakos P, Lal K. Computer-assisted design/computer-assisted manufacturing zirconia implant fixed complete prostheses: clinical results and technical complications up to 4 years of function. Clin Oral Implants Res. 2013 Jun;24(6):659-65. doi: 10.1111/j.1600-0501.2012.02447.x. Epub 2012 Mar 13. PMID 22413889
- [Background] Papaspyridakos P, Lal K. Immediate loading of the maxilla with prefabricated interim prosthesis using interactive planning software, and CAD/CAM rehabilitation with definitive zirconia prosthesis: 2-year clinical follow-up. J Esthet Restor Dent. 2010 Aug;22(4):223-32. doi: 10.1111/j.1708-8240.2010.00343.x. PMID 20690950
- [Background] Piconi C, Maccauro G. Zirconia as a ceramic biomaterial. Biomaterials. 1999 Jan;20(1):1-25. doi: 10.1016/s0142-9612(98)00010-6. PMID 9916767
- [Background] Pozzi A, Holst S, Fabbri G, Tallarico M. Clinical reliability of CAD/CAM cross-arch zirconia bridges on immediately loaded implants placed with computer-assisted/template-guided surgery: a retrospective study with a follow-up between 3 and 5 years. Clin Implant Dent Relat Res. 2015 Jan;17 Suppl 1:e86-96. doi: 10.1111/cid.12132. Epub 2013 Aug 5. PMID 23910539
- [Background] Purcell BA, McGlumphy EA, Holloway JA, Beck FM. Prosthetic complications in mandibular metal-resin implant-fixed complete dental prostheses: a 5- to 9-year analysis. Int J Oral Maxillofac Implants. 2008 Sep-Oct;23(5):847-57. PMID 19014154
- [Background] Rimondini L, Cerroni L, Carrassi A, Torricelli P. Bacterial colonization of zirconia ceramic surfaces: an in vitro and in vivo study. Int J Oral Maxillofac Implants. 2002 Nov-Dec;17(6):793-8. PMID 12507238
- [Background] Rojas-Vizcaya F. Full zirconia fixed detachable implant-retained restorations manufactured from monolithic zirconia: clinical report after two years in service. J Prosthodont. 2011 Oct;20(7):570-6. doi: 10.1111/j.1532-849X.2011.00784.x. PMID 22003832
- [Background] Slade GD. Derivation and validation of a short-form oral health impact profile. Community Dent Oral Epidemiol. 1997 Aug;25(4):284-90. doi: 10.1111/j.1600-0528.1997.tb00941.x. PMID 9332805
- [Background] Slade GD, Akinkugbe AA, Sanders AE. Projections of U.S. Edentulism prevalence following 5 decades of decline. J Dent Res. 2014 Oct;93(10):959-65. doi: 10.1177/0022034514546165. Epub 2014 Aug 21. PMID 25146182
- [Background] Thalji GN, Cooper LF. Implant-supported fixed dental rehabilitation with monolithic zirconia: a clinical case report. J Esthet Restor Dent. 2014 Mar-Apr;26(2):88-96. doi: 10.1111/jerd.12078. Epub 2014 Jan 2. PMID 24382100
- [Background] Turkyilmaz I, Company AM, McGlumphy EA. Should edentulous patients be constrained to removable complete dentures? The use of dental implants to improve the quality of life for edentulous patients. Gerodontology. 2010 Mar;27(1):3-10. doi: 10.1111/j.1741-2358.2009.00294.x. Epub 2009 Mar 8. PMID 19291086
- [Background] Venezia P, Torsello F, Cavalcanti R, D'Amato S. Retrospective analysis of 26 complete-arch implant-supported monolithic zirconia prostheses with feldspathic porcelain veneering limited to the facial surface. J Prosthet Dent. 2015 Oct;114(4):506-12. doi: 10.1016/j.prosdent.2015.02.010. Epub 2015 Jun 5. PMID 25979446